CLINICAL TRIAL: NCT02809391
Title: Orthotics and Parkinson's Disease: The Acute and Long-term Effects of Increased Somatosensory Feedback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Kelly Robb, master's student, Wilfrid Laurier University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KR_POG
Record Dates: First submitted 2016-06-13; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson Disease
Keywords: Postural Balance; Gait; Foot Orthotic; Proprioception; Somatosensory
MeSH Terms: conditions — Parkinson Disease | interventions — Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orthotic (Active Comparator): Recruited participants will be asked to wear the customizable foot orthotic, from baseline testing to a follow-up at 6 weeks post-baseline. Outcome measures at 6 weeks will be compared to those at baseline.
  Interventions: Device: Orthotics alone
- Orthotic+Textured Top Cover (Active Comparator): At 6 weeks post-baseline, participants will received a different orthotic which has a textured material used as its top cover. Testing at 6 weeks post-baseline will determine if acute changes occur as a result of wearing the orthotic with textured top cover. Testing at 12 weeks post-baseline will determine if long-term changes occur as a result of the orthotic with textured top cover.
  Interventions: Device: Orthotics+textured top cover

INTERVENTIONS:
Device: Orthotics alone — The sole thin sport orthotic will be heat moulded to participants footwear. A top cover will be used of similar cushioning thickness and durometer properties as the orthotics+texture intervention.
  Other Names: Sole thin sport orthotic
  Arms: Orthotic
Device: Orthotics+textured top cover — The sole thin sport orthotic will be heat moulded to participants footwear. A textured material will be used as the orthotic top cover in this intervention.
  Other Names: Sole thin sport orthotics with textured top cover
  Arms: Orthotic+Textured Top Cover

SUMMARY:
The purpose of this study is to increase clinical knowledge of the relationship between increased plantar sensory information and orthotics in a Parkinsonian gait. The objectives of this study are to determine if orthotics, with and without a textured top cover, can alter muscle activation, gait parameters, balance, functional mobility, and decrease fall risks in Parkinson's participants.

DETAILED DESCRIPTION:
The purpose of this study is to increase clinical knowledge of the relationship between increased plantar sensory information and orthotics in a Parkinsonian gait. Observing gait parameters and muscle activation changes, in orthotics with and without a textured top cover, provides an increased understanding of conservative treatment options available to the Parkinson's population. It is hypothesized that balance and functional mobility in Parkinson's Disease (PD) patients will increase, while decreasing fall risks, when wearing both types of orthotics. Larger improvements are expected with the orthotics with a textured top cover, thus increasing plantar sensory feedback. Male and female participants, aged 55-75, with a diagnosis of idiopathic Parkinson's disease can participate in the study. Two types of orthotic design will be examined: 1) Customizable over-the-counter orthotics and 2) Customizable over-the-counter orthotics with a textured top cover. Five different assessments will be performed during three different testing sessions: 1) baseline testing; 2) 6-weeks post-baseline; and 3) 12-weeks post-baseline. The administered assessments include: 1) Static balance, double limb stance; 2) The Berg Balance Scale (BBS); 3) Timed Up and Go (TUG), 4) Functional Gait Assessment (FGA); and 5) Walking task.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with idiopathic Parkinson' disease

Exclusion Criteria: A pre-screening questionnaire will assess the following:

* peripheral neuropathy, vestibular concerns, cognitive impairment, severe arthritic conditions, or other conflicting medical conditions
* deep brain stimulation
* currently wearing orthotics, or previously worn in the last two years
* decreased plantar sole sensation
* requires the ability to walk 10m unassisted

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change in Postural Sway during Static Stance | 6 weeks and 12 weeks post-baseline
  Static balance will be measured by the amount of postural sway in both the medio-lateral (ML) and antero-posterior (AP) directions. Participants will be asked to stand, without movement, on the pressure platform for 2 minutes. The force platform will measure the amount of spatio-temporal firing patterns from the sensory afferents in the plantar surface of participant's feet. Secondly, the IRED markers placed on participants clothing, will measure the center of mass (COM) changes in relation to the base of support (BOS). An improvement in the location of the COM in relation to the BOS suggests an improvement in balance, resulting from increased cutaneous sensation from the textured material.
Change in Dynamic Balance, using the Berg Balance Scale, Timed Up and Go, and the Functional Gait Assessment | 6 weeks and 12 weeks post-baseline
  Improvements in dynamic balance and postural stability will be defined by score improvements on the BBS, TUG, and FGA assessments. Furthermore, plantar pressure changes will be recorded during the walking task to determine if simple changes in top cover design can alter the cutaneous information from the plantar surface of the foot. Observations will be made of the plantar pressure distribution changes between the orthotic, with and without a textured top cover, in comparison to participants walking patterns with footwear alone.

SECONDARY OUTCOMES:
Change in Plantar Pressure Distribution | 6 weeks and 12 weeks post-baseline
  Force platform data will detail participant's plantar pressure distribution. Changes in plantar pressures will be recorded at 6-weeks and 12-weeks post-baseline. Pressure patterns can visually demonstrate the precise location of pressure changes on the plantar sole of the foot. Secondly, peak forces and increased load can be isolated to specific areas of the plantar sole of the foot, in relation to the total stance phase of the gait cycle (heel strike, midstance, forefoot load, and toe-off).
Change in Stride Length | 6 weeks and 12 weeks post-baseline
  Force platform data will be recorded for each participant. The anterior-posterior displacement of the ankle markers will be used to determine stride length, defined as the distance between heel strikes of the same limb.
Change in Stride Width | 6 weeks and 12 weeks post-baseline
  Force platform data will be recorded for each participant. Platform data and marker placement on participants will determine stride width, also known as base of gait, which is defined as the lateral distance between midlines of each foot.
Change in Single Limb Support Time | 6 weeks and 12 weeks post-baseline
  Force platform data will be recorded for each participant. Single limb support time is the duration of weight bearing, when only 1 limb is on contact with the ground. The force platform will record the duration of time a participant spends weight bearing on each limb.
Change in Walking Velocity | 6 weeks and 12 weeks post-baseline
  Walking velocity, or speed of gait, will be recoded by the force platform data.
Change in Electromyography (EMG) Activity | 6 weeks and 12 weeks post-baseline
  Muscle activity will be measured through EMG recordings of the tibialis anterior, peroneus longus, and gastrochnemius musculature. Secondly, changes in muscle activity will be observed in the orthotics alone compared to the textured top cover condition. The study will evaluate if the length, timing, and magnitude of the tibialis anterior, peroneus longus, and gastrochnemius properties altered with the use of orthotics, with and without a textured top cover, compared to footwear alone.
  EMG data analysis will be isolated to the stance phase of gait for each of the three muscles. The time of muscle onset and offset will be recorded within the stance phase. This will determine the location and total percentage of the stance phase each muscle activity occupied. The length of activation, the muscle's specific start and stop time of activation, and magnitude of activation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Robb, B.A.Kin, C Ped. (C), Principal Investigator — Wilfrid Laurier University
Locations (1):
- Wilfrid Laurier University, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenkins ME, Almeida QJ, Spaulding SJ, van Oostveen RB, Holmes JD, Johnson AM, Perry SD. Plantar cutaneous sensory stimulation improves single-limb support time, and EMG activation patterns among individuals with Parkinson's disease. Parkinsonism Relat Disord. 2009 Nov;15(9):697-702. doi: 10.1016/j.parkreldis.2009.04.004. Epub 2009 May 20. PMID 19467910
- [Background] Gross MT, Mercer VS, Lin FC. Effects of foot orthoses on balance in older adults. J Orthop Sports Phys Ther. 2012 Jul;42(7):649-57. doi: 10.2519/jospt.2012.3944. Epub 2012 Jan 25. PMID 22282317